CLINICAL TRIAL: NCT01486771
Title: A Pilot Study to Determine if Intravitreal Injections of Pegaptanib Sodium (Macugen) Given Every 12 Weeks for a Year After an Induction Phase of Three Injections Every 6 Weeks Will Reduce the Progression of Proliferative Diabetic Retinopathy in Patients Without Significant Vitreous Hemorrhage in Comparison to Treatment With Retinal Photocoagulation Alone and After an Induction Phase
Brief Title: Macugen for Proliferative Diabetic Retinopathy Study With Extended Dosing (M-PDRS ED)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Valley Retina Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Victor H. Gonzalez, MD, Principal Investigator, Valley Retina Institute
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MPDRS-ED
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2011-12-06 (Estimated); Status verified 2011-12

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — pegaptanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IV Macugen Q6 (Experimental): Will receive 3 intravitreal pegaptanib injections at 6-week intervals, then 3 additional injections at 12-week intervals
  Interventions: Drug: Macugen ® (pegaptanib sodium)
- IV Mac Q6 Arm (Experimental): Will Selective Laser Photocoagulation after 3 intravitreal pegaptanib injections
  Interventions: Drug: Macugen ® (pegaptanib sodium)
- Pan Retinal Photocoagulation (Experimental): Will act as the control group, thus subjects in this group will receive standard PRP (modified ETDRS protocol)
  Interventions: Drug: Macugen ® (pegaptanib sodium)

INTERVENTIONS:
Drug: Macugen ® (pegaptanib sodium) — Patients assigned to either IV Mac Q6Arm will receive a total of 3 intravitreal pegaptanib sodium injections administered at 6-week intervals beginning on Day 0 and ending at Week 12. The group will then receive an intravitreal injection every 12 weeks.
  Patients assigned to IV Mac Q6Arm will receive a total of 3 intravitreal pegaptanib sodium injections administered at 6-week intervals beginning on Day 0 and ending at Week 12. After the third injection subjects in this group will receive Selective Laser Photocoagulation at Week 18.
  Patients assigned to Panretinal Photocoagulation will act as the control group. Subjects in this group will receive standard Panretinal Photocoagulation using a modified ETDRS protocol.
  All intravitreal study injections will consist of 0.3 milligrams (mg) of pegaptanib sodium delivered by intravitreal injection.

SUMMARY:
Intravitreal injections of pegaptanib will induce the regression of Proliferative Diabetic Retinopathy (PDR) and reduce the need for retinal photocoagulation.

DETAILED DESCRIPTION:
Primary Objective:

To further establish the efficacy of intravitreal pegaptanib injections in the regression of retinal neovascularization secondary to high-risk PDR, as compared to standard panretinal photocoagulation (PRP)

Secondary Objective:

To maintain the regression of PDR after the induction phase with intravitreal pegaptanib injections administered at 12-week intervals, as compared to standard PRP

To maintain the regression of PDR after the induction phase with retinal photocoagulation applied to areas of ischemia (Selective Laser Photocoagulation), as compared to standard PRP

To evaluate the rate of recurrence of neovascularization after 6 intravitreal pegaptanib injections

To determine if intravitreal pegaptanib will reduce the area and/or volume of concomitant diabetic macular edema, as assessed by leakage on fluorescein angiography (FA) and/or optical coherence tomography (OCT)

To determine if intravitreal pegaptanib injections maintain or reduce the loss of best-corrected visual acuity

ELIGIBILITY:
Inclusion Criteria:

1. Eligible eyes will have active PDR with high risk characteristics (HRC) as defined by the DRS. All eyes must meet at least one or both of the following criteria:

   * Mild neovascularization of the disc (NVD) of at least 1/4 to 1/3 disc area as shown in standard photograph 10A of the DRS.
   * Moderate neovascularization of the retina elsewhere (NVE) of at least 1/2 disc area as shown in standard photograph 7 of the DRS.
2. ETDRS visual acuity score greater than or equal to 24 letters (approximately 20/320) and less than or equal to 85 letters (approximately 20/20) by the ETDRS visual acuity protocol at the screening visit.
3. Eyes with mild pre-retinal hemorrhage (PRH) or mild vitreous hemorrhage (VH) that does not interfere with clear visualization of the macula and optic disc are eligible for this study.
4. Evaluating physician believes that PRP can be safely withheld for 3 weeks.

Exclusion Criteria:

1. Presence of moderate or dense PRH or VH that prevents clear visualization of the macula and/or optic disc.
2. Presence of either:

   * significant epiretinal membranes involving the macula, OR
   * proliferative diabetic membranes along the major retinal arcades that are extensive enough to cause either:

     * significant vitreomacular traction, OR
     * significant impairment in visual acuity.
3. Presence of any tractional retinal detachment.
4. Severe ischemia involving the foveal avascular zone as determined by fluorescein angiography performed at the initial screening visit.
5. Significant media opacity (due to cornea, anterior chamber, or lens) precluding clear visualization of the macula or optic disc.
6. Presence of neovascular glaucoma with or without hyphema.
7. Previous treatment with intravitreal steroid injections in the study eye within 6 months of baseline.
8. Previous treatment with peribulbar steroid injections in the study eye within 90 days of baseline
9. Previous PRP laser treatment in the study eye within 90 days of baseline visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-11; Primary Completion 2013-08 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Establish efficacy of intravitreal pegaptanib sodium injections in causing regression of high risk proliferative diabetic retinopathy as compared to panretinal photocoagulation | 54 weeks
  To assess the efficacy of intravitreal pegaptanib sodium injections in inducing regression of high risk PDR (as determined by percentage of eyes without treatment failure) using standard panretinal photocoagulation (PRP) as the control arm. Treatment failure is defined as:
  * Development of increased NVD and/or NVE
  * NVD and/or NVE that is not regressed at least 50% compared to the baseline amount within 3 weeks
  * Development of significant vitreous hemorrhage that is sufficient in quantity to obscure visualization of the entire macula, optic disc, and the major temporal arcade vessels

SECONDARY OUTCOMES:
Establish the efficacy of intravitreal pegaptanib injections in preventing the loss of best corrected visual acuity | 54 weeks
  To determine if intravitreal pegaptanib sodium injections maintain or reduce the loss of best-corrected visual acuity as measured by comparing the percentages of patients that lost 3 or more lines on ETDRS chart in the study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Victor H. Gonzalez, MD, Principal Investigator — Valley Retina Insitute
Locations (1):
- Valley Retina Insitute, PA, McAllen, Texas, United States